CLINICAL TRIAL: NCT06671171
Title: Wearable Assessment of Thoracic, Cardiac Health and Exercise Performance Trial
Acronym: WATCH-X
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Chun Ka, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: WATCH-X; HKU / HA HKW IRB (Other: HKU / HA HKW IRB)
Record Dates: First submitted 2024-10-24; First posted 2024-11-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-10

CONDITIONS: Congenital Heart Disease; Pulmonary Hypertension; Heart Failure; Coronary Artery Disease
Keywords: congenital heart disease; pulmonary hypertension; heart failure; coronary artery disease; athletes; smartwatch
MeSH Terms: conditions — Heart Defects, Congenital; Hypertension, Pulmonary; Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- WatchX: Participants will wear the investigational smartwatch (Apple Watch Series 9) concurrently for pre- and post-SaO2 and VO2max assessment during cardiopulmonary exercise test at Visit 1.
  Through one-week study period, participants will record their oxygen saturation data collected by the smartwatch once daily in a provided log, preferably in the morning after waking and before any strenuous activity.
  At Visit 2, participants will walk for a 6-Minute walk test and wear the investigational smartwatch (Apple Watch Series 9) concurrently for pre- and post-SaO2 and VO2max assessment during assessment.
  Interventions: Device: Apple Watch Series 9

INTERVENTIONS:
Device: Apple Watch Series 9 — Participants will wear Apple Watch Series 9 during cardiopulmonary exercise test (in Visit 1), 1-week study period and 6-Minute walk distance test (in Visit 2) to have assessment of maximal oxygen uptake and pre- and post-SaO2.
  During 1-week study period, participants will measure their oxygen saturation once daily with a medical-grade pulse oximeter while wearing the smartwatch continuously.

SUMMARY:
Wearable health technology, particularly smartwatches, has revolutionized personal health monitoring by enabling continuous, non-invasive tracking of various physiological parameters. The potential applications of these devices in cardiology are extensive, but it is crucial to validate their accuracy against established medical-grade devices.

The Apple Watch Series 9 (Apple, USA) exemplifies the capabilities of modern smartwatches, offering a wide range of health tracking features. These include heart rate monitoring, detection of irregular heart rhythms suggestive of atrial fibrillation, electrocardiogram recording, blood oxygen level measurement, and comprehensive mobility metrics (including VO2 max, six-minute walk distance, walking speed, step length, double support time, and walking asymmetry). Many of these parameters are highly relevant for cardiovascular patients, potentially aiding in disease progression monitoring and adverse event prediction. However, there is a lack of comprehensive validation studies for these devices in specific cardiovascular disease populations.

This investigator-initiated prospective observational study involving 50-100 participants that aims to validate smartwatchbased assessments using medical-grade devices and techniques. The study will focus on adult patients with congenital heart disease, pulmonary hypertension, heart failure, and coronary artery disease, as well as athletes undergoing cardiovascular assessment. By comparing smartwatch data with established clinical measurements, the investigators seek to determine the reliability and potential clinical utility of these wearable devices in diverse cardiovascular contexts. This research will help bridge the gap between consumer-grade wearable technology and clinical practice in cardiology.

DETAILED DESCRIPTION:
Trial participants from Queen Mary Hospital and the University of Hong Kong will be recruited. Potential participants will be contacted and provided with a detailed explanation of the study, including its purpose, procedures, risks, and benefits. Written informed consent will be obtained from all participants before enrolment. This process involves providing individuals with the informed consent document, allowing time for review and questions, and obtaining their signature if they agree to participate. Participants will receive a copy of the signed consent form for their records.

At Visit 1, Comprehensive demographic and clinical data will be collected from each participant, Clinical Management System (CMS), Electronic Patient Record (ePR), and Clinical Data Analysis and Reporting System (CDARS) of the Hospital Authority in Hong Kong. This will include age, sex, height, weight, body mass index, and detailed medical history focusing on cardiovascular conditions. Information about current medications and smoking status will also be recorded. Additionally, participants will undergo a baseline clinical examination, including blood pressure measurement, heart rate, and a 12-lead electrocardiogram.

Participants will undergo a conventional cardiopulmonary exercise test (CPX) to determine their maximal oxygen uptake (VO2max) at Visit 1. This test will be conducted in a controlled clinical setting under the supervision of cardiologists. Participants will exercise on a treadmill while their respiratory gas exchange is measured using a metabolic cart. The exercise intensity will be gradually increased until the participant reaches volitional exhaustion or predetermined safety criteria are met. The highest oxygen uptake value achieved during the test will be recorded as the VO2max. Participant will concurrently be wearing the investigational smartwatch for pre- and post-SaO2 and VO2max assessment. This gold-standard measurement will serve as the reference for validating the smartwatch's continuous VO2max estimation.

The 6-minute walk distance will be assessed in a hospital setting at Visit 2 under the supervision of a research staff. Participants will be instructed to walk as far as possible in six minutes along a predetermined course, typically a straight hallway. The total distance walked will be measured and recorded. During the test, the research nurse will monitor the participant's heart rate, blood oxygen saturation, and perceived exertion at regular intervals. Participant will concurrently be wearing the investigational smartwatch for pre- and post SaO2 and VO2max assessment.

Participants will be provided with a medical-grade pulse oximeter for home use. They will be instructed to measure their oxygen saturation once daily throughout the one-week study period. Measurements should be taken at approximately the same time each day, preferably in the morning after waking and before any strenuous activity. Participants will record their oxygen saturation readings in a provided log. These daily measurements will serve as reference points for validating the continuous oxygen saturation data collected by the smartwatch.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 70 years old
* Ability to provide informed consent
* History of the following cardiovascular conditions
* Adult congenital heart disease
* Pulmonary hypertension
* Heart failure
* Coronary artery disease
* Athletes undergoing cardiovascular assessment

Exclusion Criteria:

* Contraindication for undergoing physical exertion including cardio-pulmonary exercise testing (CPX) and 6-minute walk test (6MWT)
* Pregnancy
* Known allergy to components of the investigational product

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with congenital heart disease, pulmonary hypertension, heart failure, and coronary artery disease, as well as athletes undergoing cardiovascular assessment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2 max, in ml/min/kg) | During treadmill exercise in the day of recruitment and concurrently baseline assessment (Visit 1/ Week 1)
  VO2 max (ml/min/kg) concurrently measured with a medical-grade device and a smartwatch during treadmill exercise as assessed during treadmill exercise

SECONDARY OUTCOMES:
Correlation between VO2 max (ml/min/kg) obtained using medical-grade device and smartwatch | From enrollment to end of follow up at Visit 2(Week 2)
  VO2 max (ml/min/kg) obtained using medical-grade device and smartwatch during supervised treadmill exercise, supervised 6-minute walk test and mean and max value during other exercise
Correlation between SaO2 (%) obtained using medical-grade device and smartwatch | From enrollment to end of follow up at Visit 2(Week 2)
  SaO2 (%) obtained using medical-grade device and smartwatch during supervised treadmill exercise, supervised 6-minute walk test and during other exercise in the follow up period.
SaO2 (%) measured by the smartwatch | From enrollment to end of follow up at Visit 2(Week 2)
  SaO2 (%) measured by the smartwatch from enrollment to end of follow up period
SaO2 (%) in participants with severe disease and participants with mild disease | From enrollment to end of follow up at Visit 2(Week 2)
  SaO2 (%) in participants with severe versus mild disease from enrollment to end of follow up period
Novel markers or patterns | From enrollment to end of follow up at Visit 2(Week 2)
  Novel markers or patterns indicative of disease severity or predictive of adverse events as assessed from enrollment to end of follow up period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine Queen Marry Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guo Y, Wang H, Zhang H, Liu T, Liang Z, Xia Y, Yan L, Xing Y, Shi H, Li S, Liu Y, Liu F, Feng M, Chen Y, Lip GYH; MAFA II Investigators. Mobile Photoplethysmographic Technology to Detect Atrial Fibrillation. J Am Coll Cardiol. 2019 Nov 12;74(19):2365-2375. doi: 10.1016/j.jacc.2019.08.019. Epub 2019 Sep 2. PMID 31487545
- [Background] Chan PH, Wong CK, Poh YC, Pun L, Leung WW, Wong YF, Wong MM, Poh MZ, Chu DW, Siu CW. Diagnostic Performance of a Smartphone-Based Photoplethysmographic Application for Atrial Fibrillation Screening in a Primary Care Setting. J Am Heart Assoc. 2016 Jul 21;5(7):e003428. doi: 10.1161/JAHA.116.003428. PMID 27444506
- [Background] Wong CK, Lau YM, Lui HW, Chan WF, San WC, Zhou M, Cheng Y, Huang D, Lai WH, Lau YM, Siu CW. Automatic detection of cardiac conditions from photos of electrocardiogram captured by smartphones. Heart. 2024 Aug 14;110(17):1074-1082. doi: 10.1136/heartjnl-2023-323822. PMID 38768982
- [Background] Mannhart D, Lischer M, Knecht S, du Fay de Lavallaz J, Strebel I, Serban T, Vogeli D, Schaer B, Osswald S, Mueller C, Kuhne M, Sticherling C, Badertscher P. Clinical Validation of 5 Direct-to-Consumer Wearable Smart Devices to Detect Atrial Fibrillation: BASEL Wearable Study. JACC Clin Electrophysiol. 2023 Feb;9(2):232-242. doi: 10.1016/j.jacep.2022.09.011. Epub 2023 Jan 18. PMID 36858690
- [Background] Perez MV, Mahaffey KW, Hedlin H, Rumsfeld JS, Garcia A, Ferris T, Balasubramanian V, Russo AM, Rajmane A, Cheung L, Hung G, Lee J, Kowey P, Talati N, Nag D, Gummidipundi SE, Beatty A, Hills MT, Desai S, Granger CB, Desai M, Turakhia MP; Apple Heart Study Investigators. Large-Scale Assessment of a Smartwatch to Identify Atrial Fibrillation. N Engl J Med. 2019 Nov 14;381(20):1909-1917. doi: 10.1056/NEJMoa1901183. PMID 31722151
- [Background] Wong CK, Un KC, Zhou M, Cheng Y, Lau YM, Shea PC, Lui HW, Zuo ML, Yin LX, Chan EW, Wong ICK, Sin SWC, Yeung PPN, Chen H, Wibowo S, Wei TLN, Lee SM, Chow A, Tong RCF, Hai J, Tam FCC, Siu CW. Daily ambulatory remote monitoring system for drug escalation in chronic heart failure with reduced ejection fraction: pilot phase of DAVID-HF study. Eur Heart J Digit Health. 2022 May 7;3(2):284-295. doi: 10.1093/ehjdh/ztac024. eCollection 2022 Jun. PMID 36713022